CLINICAL TRIAL: NCT06892379
Title: A Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of HS-20110 in Participants With Advanced Solid Tumors
Brief Title: A Study of HS-20110 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HS-20110-101
Record Dates: First submitted 2025-02-24; First posted 2025-03-24 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HS-20110 (Phase Ia：Dose escalation ) (Experimental)
  Interventions: Drug: HS-20110 (Phase Ia：Dose escalation )
- HS-20110 (Phase 1b Dose expansion) (Experimental)
  Interventions: Drug: HS-20110 (Phase Ib:Dose expansion )

INTERVENTIONS:
Drug: HS-20110 (Phase Ia：Dose escalation ) — HS-20110 for IV infusion of various dose strengths administered in 21 day dosing cycles
  Arms: HS-20110 (Phase Ia：Dose escalation )
Drug: HS-20110 (Phase Ib:Dose expansion ) — The recommended dose from the dose-escalation stage and other potential doses will be further explored
  Arms: HS-20110 (Phase 1b Dose expansion)

SUMMARY:
This is an open-label, multicenter study to evaluate the safety and tolerability of HS-20110 in participants with advanced solid malignant tumors

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, aged ≥ 18 years.
2. Participants with pathologically (histologically or cytologically) confirmed advanced solid tumors.
3. Participants have at least 1 target lesion other than CNS lesions according to RECIST 1.1.

Exclusion Criteria:

1. Participants have received or are receiving the following treatment:

   1. Drug therapy targeting CDH17 (such as small molecule targeted drugs, monoclonal antibodies, bispecific antibodies, antibody-drug conjugates, or chimeric antigen receptor T cells).
   2. Anti-tumor drugs within 14 days prior to the first dose of study treatment; any other IMPs or macromolecular anti-tumor drugs within 28 days prior to the first dose of study treatment.
   3. Local radiotherapy within 2 weeks prior to the first dose of study treatment; irradiation of more than 30% of bone marrow or extensive radiotherapy within 4 weeks prior to the first dose of study treatment.
   4. Major surgery within 4 weeks prior to the first dose of study treatment.
   5. Participants previously treated with drugs that are moderate to strong inhibitors or moderate to strong inducers of cytochrome P450 (CYP) 3A4, strong inhibitors or strong inducers of CYP2D6, P-glycoprotein (P-gp), breast cancer resistance protein (BCRP) or drugs with a narrow therapeutic range that are sensitive substrates of P-gp or BCRP within 7 days prior to the first dose of the IMP. Participants who need to receive these drugs during the study period should also be excluded.
   6. Current use of drugs known to prolong the QT interval or that may cause torsade de pointes. Participants who need to receive these drugs during the study period should also be excluded.
   7. Live vaccine or live-attenuated vaccine within 28 weeks prior to the first dose.
2. Participants who have any Grade ≥ 2 residual toxicity according to Common Terminology Criteria for Adverse Events (CTCAE, version 5.0) from prior therapies (except alopecia and residual neurotoxicity).
3. Inadequate bone marrow reserve or hepatic and renal functions.
4. Participants with a history of severe allergy (such as anaphylactic shock), previous severe infusion reactions, or allergy to recombinant human or murine proteins.
5. Participants who are allergic to any component of HS-20110.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) or maximum applicable dose (MAD) | From day 1 to one months after the last dose in Phase 1a
Objective response rate (ORR) as per RECIST v1.1 | From screening to 2 months after the last dose

SECONDARY OUTCOMES:
Incidence of adverse events (AEs), serious adverse events (SAEs), AEs leading to dose modification or permanent discontinuation, and specific laboratory abnormalities | From the first dose until 90 days after the last dose
Objective response rate (ORR), disease control rate (DCR), duration of response (DoR), and progression-free survival (PFS) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1; overall survival (OS) | From screening to up to 3 years after last dose
Incidence of anti-HS-20110 antibody (ADA) | From the first dose until 90 days after the last dose
Drug concentrations of the three components of HS-20110 (including antibody-drug conjugates, total antibody, and payload) | From the first dose until 90 days after the last dose

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - BRCR Medical Center INC, Tamarac, Florida
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- SUN YAT-SEN University Cancer Center, Guangzhou, Guangdong, China